CLINICAL TRIAL: NCT06735755
Title: A Phase 1/2, Dose-Exploration Study to Evaluate the Safety and Efficacy of BEAM-301 in Patients With Glycogen Storage Disease Type Ia (GSDIa) Homozygous or Compound Heterozygous for the G6PC1 c.247C>T (p.R83C) Variant
Brief Title: A Phase 1/2, Dose-Exploration Study to Evaluate the Safety and Efficacy of BEAM-301 in Patients With Glycogen Storage Disease Type Ia (GSDIa)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beam Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BTX-301-001
Record Dates: First submitted 2024-12-06; First posted 2024-12-16 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Glycogen Storage Disease Type Ia
Keywords: GSDIa; GSD1a
MeSH Terms: conditions — Hepatorenal form of glycogen storage disease

STUDY DESIGN:
Intervention Model Description: up to 4 planned, single-ascending-dose, dose-exploration cohorts
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BEAM-301 (Experimental): BEAM-301 consists of adenine base editor messenger ribonucleic acid (mRNA) and single guide ribonucleic acid (gRNA) formulated in lipid nanoparticles (LNPs) for intravenous (IV) administration.
  Interventions: Drug: BEAM-301: Single dose of BEAM-301 administered by IV

INTERVENTIONS:
Drug: BEAM-301: Single dose of BEAM-301 administered by IV — BEAM-301 is designed to correct the G6PC1 c.247C>T allele via an A:T-to-G:C base-pair substitution, resulting in restoration of G6Pase-α catalytic activity.

SUMMARY:
This is a Phase 1/2, multicenter, open-label, single-ascending-dose study to evaluate the safety, tolerability, and efficacy of BEAM-301 in adult patients with GSDIa homozygous or compound heterozygous for the G6PC1 c.247C>T (p.R83C) variant and to determine the optimal biological dose.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age ≥18 years of age at the time of consent.
2. Diagnosis of GSDIa and homozygous or compound heterozygous for the G6PC1 c.247C>T (p.R83C) variant (confirmed by genetic testing).
3. History of at least 1 episode of hypoglycemia <60 mg/dL within the 2 years prior to signing the ICF.

Exclusion Criteria:

1. Liver transplant recipient/on waiting list for liver transplant or known history of liver cirrhosis.
2. Presence of liver adenoma >5 cm in size based on liver MRI or liver ultrasound performed at screening or within 6 months prior to screening.
3. Presence of liver adenoma >3 cm and ≤5 cm with a documented annual growth rate of ≥0.5 cm per year.
4. Have aspartate transaminase or alanine transaminase >upper limit of normal (ULN).
5. Total bilirubin levels >ULN; if documented Gilbert's Syndrome, total bilirubin >2 × ULN.
6. Previous treatment with any cell-, gene-, or viral vector-derived therapy Hospitalization for management of hypoglycemia within 4 weeks prior to signing the ICF.
7. Have triglycerides >1000 mg/dL or a history of pancreatitis or a history of acute pancreatitis within 5 years that does not have a known and corrected etiology (eg, cholecystectomy for gallstone pancreatitis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BEAM-301 in patients with GSDIa with a G6PC1 c.247C>T (p.R83C) variant by measuring incidence of treatment-emergent adverse events (TEAEs) including serious adverse events (SAEs) and dose-limiting toxicities (DL | BEAM-301 administration through month 24

SECONDARY OUTCOMES:
Absolute and change from baseline in time to hypoglycemia or metabolic decompensation during a controlled fasting challenge | Baseline to month 24
Changes from baseline in starch supplementation dose | Baseline to month 24
Level of serum glucose and metabolic parameters (lipid profile and uric acid) over time | Baseline to month 24
BEAM-301 PK parameters (Cmax) | Baseline to month 24
BEAM-301 PK parameters (AUC) | Baseline to month 24
BEAM-301 PK parameters (half-life) | Baseline to month 24

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Clinical Study Site, Orange, California
  - Clinical Study Site, Farmington, Connecticut
  - Clinical Study Site, Houston, Texas